CLINICAL TRIAL: NCT03243409
Title: Perioperative Complications in Proximal Humeral Fractures Treated With Reversed Shoulder Arthroplasties
Brief Title: Perioperative Complications in Reversed Shoulder Arthroplasties
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-HUM-2017-51
Record Dates: First submitted 2017-07-31; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Proximal Humeral Fracture
Keywords: reversed shoulder arthroplasties; clinical complications; complex proximal humeral fractures
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective observational study of reversed shoulder arthroplasties by proximal humeral fracture. Analysis of preoperative risk factors as well as minor and major complications at the first week, 90 days and 1 year.

DETAILED DESCRIPTION:
The study is a multicenter retrospective observational study (3 centers). Data are collected from 105 patients over 65 years-old undergoing reversed shoulder arthroplasties by proximal humerus fractures, in 3 or 4 parts.

Patient information is obtained from the clinical records in their usual preoperative assessment, and follow-up on the usual routine checks, at the first week, 90 days and 1 year.

Minor and major complications rates are evaluated according to preoperative risk (ASA), underlying diseases and according to anticoagulant / antiaggregant treatments.

Likewise, transfusion rates related to ASA, as well as length of hospital stay related to it.

ELIGIBILITY:
Inclusion Criteria:

* Complex( 3- or 4-part) humerus fractures undergoing reversed shoulder arthroplasties.

Exclusion Criteria:

* No exclusion criteria

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients undergoing reversed shoulder arthroplasties owing to three or four parts fractures of the proximal humerus
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2017-08-31 (Estimated); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients affected by minor complications according to preoperative risk (ASA) in reversed shoulder arthroplasties due to complex proximal humeral fractures. | First week after surgery
  Minor complications are medical complications, which usually don't affect to the functional outcome of arthroplasties
Number of patients affected by minor complications according to preoperative risk (ASA) in reversed shoulder arthroplasties due to complex proximal humeral fractures. | 90 days after surgery
  Minor complications are medical complications, which usually don't affect to the functional outcome of arthroplasties
Number of patients affected by minor complications according to preoperative risk (ASA) in reversed shoulder arthroplasties due to complex proximal humeral fractures. | 1 year after surgery
  Minor complications are medical complications, which usually don't affect to the functional outcome of arthroplasties
Number of patients affected by major complications according to preoperative risk (ASA) in reversed shoulder arthroplasties due to complex proximal humeral fractures. | First week after surgery
  Major complications are surgical complications( dislocation, periprosthetic fracture, infection) which usually affect to the functional outcome and can lead to a revision surgery
Number of patients affected by major complications according to preoperative risk (ASA) in reversed shoulder arthroplasties due to complex proximal humeral fractures. | 90 days after surgery
  Major complications are surgical complications( dislocation, periprosthetic fracture, infection) which usually affect to the functional outcome and can lead to a revision surgery
Number of patients affected by major complications according to preoperative risk (ASA) in reversed shoulder arthroplasties due to complex proximal humeral fractures. | 1 year after surgery
  Major complications are surgical complications( dislocation, periprosthetic fracture, infection) which usually affect to the functional outcome and can lead to a revision surgery

SECONDARY OUTCOMES:
Number of patients affected by minor complications after surgery, according to underlying disease | First week after surgery
  Underlying diseases group: cardiovascular, neurological, rheumatic, psychiatric, neoplasic.
Number of patients with cardiovascular diseases affected by minor complications after surgery | 90 days after surgery
  Underlying diseases group: cardiovascular, neurological, rheumatic, psychiatric, neoplasic.
Number of patients with cardiovascular diseases affected by minor complications after surgery | 1 year after surgery
  Underlying diseases group: cardiovascular, neurological, rheumatic, psychiatric, neoplasic.
Number of patients with cardiovascular diseases affected by major complications after surgery | First week after surgery
  Underlying diseases group: cardiovascular, neurological, rheumatic, psychiatric, neoplasic.
Number of patients with cardiovascular diseases affected by major complications after surgery | 90 days after surgery
  Underlying diseases group: cardiovascular, neurological, rheumatic, psychiatric, neoplasic.
Number of patients with cardiovascular diseases affected by major complications after surgery | 1 year after surgery
  Underlying diseases group: cardiovascular, neurological, rheumatic, psychiatric, neoplasic.
Number of patients undergoing anticoagulant treatment with minor complications | First week after surgery
  Previous acenocoumarol treatment
Number of patients undergoing anticoagulant treatment with major complications | First week after surgery
  Previous acenocoumarol treatment
Number of patients undergoing anticoagulant treatment with minor complications | 90 days after surgery
  Previous acenocoumarol treatment
Number of patients undergoing anticoagulant treatment with major complications | 90 days after surgery
  Previous acenocoumarol treatment
Number of patients undergoing antiplatelet treatment with minor complications | First week after surgery
  Previous Acetylsalicylic acid (Aspirin), triflusal, ticlopidine, clopidogrel or prasugrel
Number of patients undergoing antiplatelet treatment with major complications | First week after surgery
  Previous Acetylsalicylic acid (Aspirin), triflusal, ticlopidine, clopidogrel or prasugrel
Number of patients undergoing antiplatelet treatment with minor complications | 90 days after surgery
  Previous Acetylsalicylic acid (Aspirin), triflusal, ticlopidine, clopidogrel or prasugrel
Number of patients undergoing antiplatelet treatment with major complications | 90 days after surgery
  Previous Acetylsalicylic acid (Aspirin), triflusal, ticlopidine, clopidogrel or prasugrel
Transfusion rates according to the preoperative ASA group | 1 week after surgery
  Number of transfusion requirement.
Length of hospital stay according to the preoperative ASA group | 1 week after surgery
  Length from the surgical intervention according to ASA risk

CONTACTS AND LOCATIONS:
Overall Officials: Carles Torrens Canovas, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrel JR, Trinh TQ, Fischer RA. Reverse total shoulder arthroplasty versus hemiarthroplasty for proximal humeral fractures: a systematic review. J Orthop Trauma. 2015 Jan;29(1):60-8. doi: 10.1097/BOT.0000000000000224. PMID 25186842
- [Background] Boileau P, Winter M, Cikes A, Han Y, Carles M, Walch G, Schwartz DG. Can surgeons predict what makes a good hemiarthroplasty for fracture? J Shoulder Elbow Surg. 2013 Nov;22(11):1495-506. doi: 10.1016/j.jse.2013.04.018. Epub 2013 Jul 5. PMID 23834993
- [Background] Bufquin T, Hersan A, Hubert L, Massin P. Reverse shoulder arthroplasty for the treatment of three- and four-part fractures of the proximal humerus in the elderly: a prospective review of 43 cases with a short-term follow-up. J Bone Joint Surg Br. 2007 Apr;89(4):516-20. doi: 10.1302/0301-620X.89B4.18435. PMID 17463122
- [Background] Stanbury SJ, Voloshin I. Reverse shoulder arthroplasty for acute proximal humeral fractures in the geriatric patient: a review of the literature. Geriatr Orthop Surg Rehabil. 2011 Sep;2(5-6):181-6. doi: 10.1177/2151458511420140. PMID 23569688
- [Background] Cuff DJ, Pupello DR. Comparison of hemiarthroplasty and reverse shoulder arthroplasty for the treatment of proximal humeral fractures in elderly patients. J Bone Joint Surg Am. 2013 Nov 20;95(22):2050-5. doi: 10.2106/JBJS.L.01637. PMID 24257664
- [Background] Boyle MJ, Youn SM, Frampton CM, Ball CM. Functional outcomes of reverse shoulder arthroplasty compared with hemiarthroplasty for acute proximal humeral fractures. J Shoulder Elbow Surg. 2013 Jan;22(1):32-7. doi: 10.1016/j.jse.2012.03.006. Epub 2012 May 29. PMID 22652065
- [Background] Jones KJ, Dines DM, Gulotta L, Dines JS. Management of proximal humerus fractures utilizing reverse total shoulder arthroplasty. Curr Rev Musculoskelet Med. 2013 Mar;6(1):63-70. doi: 10.1007/s12178-013-9155-1. PMID 23334846
- [Background] Lenarz C, Shishani Y, McCrum C, Nowinski RJ, Edwards TB, Gobezie R. Is reverse shoulder arthroplasty appropriate for the treatment of fractures in the older patient? Early observations. Clin Orthop Relat Res. 2011 Dec;469(12):3324-31. doi: 10.1007/s11999-011-2055-z. PMID 21879403
- [Background] Chalmers PN, Slikker W 3rd, Mall NA, Gupta AK, Rahman Z, Enriquez D, Nicholson GP. Author reply: reverse total shoulder for acute proximal humeral fracture: comparison to open reduction-internal fixation and hemiarthroplasty. J Shoulder Elbow Surg. 2014 Sep;23(9):e222. doi: 10.1016/j.jse.2014.05.014. Epub 2014 Jul 24. No abstract available. PMID 25066822
- [Background] Acevedo DC, Vanbeek C, Lazarus MD, Williams GR, Abboud JA. Reverse shoulder arthroplasty for proximal humeral fractures: update on indications, technique, and results. J Shoulder Elbow Surg. 2014 Feb;23(2):279-89. doi: 10.1016/j.jse.2013.10.003. PMID 24418780
- [Background] Mata-Fink A, Meinke M, Jones C, Kim B, Bell JE. Reverse shoulder arthroplasty for treatment of proximal humeral fractures in older adults: a systematic review. J Shoulder Elbow Surg. 2013 Dec;22(12):1737-48. doi: 10.1016/j.jse.2013.08.021. PMID 24246529
- [Background] Sebastia-Forcada E, Cebrian-Gomez R, Lizaur-Utrilla A, Gil-Guillen V. Reverse shoulder arthroplasty versus hemiarthroplasty for acute proximal humeral fractures. A blinded, randomized, controlled, prospective study. J Shoulder Elbow Surg. 2014 Oct;23(10):1419-26. doi: 10.1016/j.jse.2014.06.035. Epub 2014 Jul 30. PMID 25086490
- [Background] Wall B, Walch G. Reverse shoulder arthroplasty for the treatment of proximal humeral fractures. Hand Clin. 2007 Nov;23(4):425-30, v-vi. doi: 10.1016/j.hcl.2007.08.002. PMID 18054669